CLINICAL TRIAL: NCT00300677
Title: Assessment Of Voriconazole Penetration Into The Brain By Fluorine-Magnetic Resonance Spectroscopy
Brief Title: To Determine The Amount Of Voriconazole In The Brain After 2 Loading Doses And 3 Maintenance Doses Over 3 Days
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: McLean Hospital. Belmont, MA. (Unknown)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A1501079
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Infections, Fungal
Keywords: Pharmacokinetics; Voriconazole; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- voriconazole (Experimental): voriconazole twice daily
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — Multiple oral doses of voriconazole at 400 mg loading twice daily followed by 200 mg maintenance twice daily
  Other Names: Vfend

SUMMARY:
To determine the amount of voriconazole in the brain after 2 loading doses and 3 maintenance doses over 3 days and compare it to the amount of voriconazole in the plasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide informed consent.
* Subjects must be willing and able to be confined at the Clinical Research Unit as required by the protocol.

Exclusion Criteria:

* Subjects with any condition affecting drug absorption.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] Henry ME, Bolo NR, Zuo CS, Villafuerte RA, Cayetano K, Glue P, Damle BD, Andrews E, Lauriat TL, Rana NS, Churchill JH, Renshaw PF. Quantification of brain voriconazole levels in healthy adults using fluorine magnetic resonance spectroscopy. Antimicrob Agents Chemother. 2013 Nov;57(11):5271-6. doi: 10.1128/AAC.00394-13. Epub 2013 Aug 12. PMID 23939898
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501079&StudyName=To%20Determine%20The%20Amount%20Of%20Voriconazole%20In%20The%20Brain%20After%202%20Loading%20Doses%20And%203%20Maintenance%20Doses%20Over%203%20Days%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male volunteers were recruited by 1 hospital center in the U.S. between March 2007 and August 2008.
Groups:
- Voriconazole: 400 mg every 12 hours on Day 1; 200 mg every 12 hours on Day 2; 200 mg on Day 3
Period: Overall Study
Arm/Group | Voriconazole
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  18-25 years | 3
  26-35 years | 6
  36-45 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentrations of Voriconazole
Description: Mean plasma voriconazole concentrations (nanograms per milliliter [ng/mL]) pre-dose (Cmin) and two hours post-dose (C2h). Plasma samples were assayed using a validated, sensitive, and specific high performance liquid chromatography/tandem mass spectrometry (HPLC-MS/MS) method.
Time Frame: Day 3: pre-dose, 2 hours post-dose
Population: Pharmacokinetic Analysis Set: subjects included in the statistical analysis of pharmacokinetic parameters had the pharmacokinetic parameter of interest. N=number of observations (non-missing concentrations).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voriconazole
Number analyzed (Participants) | 12
ng/mL
  predose (Cmin) | 839.50 (874.22)
  2 hours postdose (C2h) | 2182.33 (1190.63)
Statistical Analysis 1: Comparison: Voriconazole; Other estimated parameter represents the Day 3 pre-dose ratio of the adjusted geometric means comparing brain vs. plasma concentrations of voriconazole. Natural-log transformed concentrations of voriconazole were analyzed using a mixed-effects model to obtain the adjusted mean difference (Test-Reference) and 90% confidence interval for the difference which were exponentiated to provide estimates of the ratio of the adjusted geometric means and 90% CI for the ratio; Test type: Superiority or Other; ANOVA; Mixed-effects analysis of variance model with time, compartment, and time by compartment interaction as fixed effects and subjects as random effects; predose: ratio adjusted geometric means = 300.28, 90% CI [192.91 to 467.43] — Estimated value = ratio (%) of adjusted geometric means comparing brain (test) vs. plasma (reference) concentrations of voriconazole
Statistical Analysis 2: Comparison: Voriconazole; Other estimated parameter represents the Day 3 post-dose ratio of the adjusted geometric means comparing brain vs. plasma concentrations of voriconazole. Natural-log transformed concentrations of voriconazole were analyzed using a mixed-effects model to obtain the adjusted mean difference (Test-Reference) and 90% confidence interval for the difference which were exponentiated to provide estimates of the ratio of the adjusted geometric means and 90% CI for the ratio; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; postdose: ratio adjusted geometric means = 192.72, 90% CI [123.81 to 300.00] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Brain Concentrations of Voriconazole
Description: Mean brain concentrations (ng/mL) of voriconazole pre-dose and 2 hours post-dose measured by Fluorine (F) Magnetic Resonance Spectroscopy (F-MRS).
Time Frame: Day 3: pre-dose, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voriconazole
Number analyzed (Participants) | 12
ng/mL
  predose (Cmin) | 2090.44 (1227.88)
  2 hours postdose (C2h) | 4165.20 (1806.93)
Statistical Analysis 1: Comparison: Voriconazole; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; predose: ratio adjusted geometric means = 300.28, 90% CI [192.91 to 467.43] — Estimated value = ratio (%) of the adjusted geometric means comparing brain (test) vs. plasma (reference) concentrations of voriconazole
Statistical Analysis 2: Comparison: Voriconazole; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; postdose: ratio adjusted geometric means = 192.72, 90% CI [123.81 to 300.00] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Plasma Concentrations of N-oxide Metabolite
Description: Mean plasma concentrations of voriconazole N-oxide metabolite (ng/mL) pre-dose and 2 hours post-dose. Plasma samples were assayed using a validated, sensitive, and specific high performance liquid chromatography/tandem mass spectrometry (HPLC-MS/MS) method.
Time Frame: Day 3: pre-dose, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voriconazole
Number analyzed (Participants) | 12
ng/mL
  predose (Cmin) | 3076.67 (841.96)
  2 hours postdose (C2h) | 3665.00 (958.73)
Statistical Analysis 1: Comparison: Voriconazole; Other estimated parameter represents the Day 3 pre-dose ratio of the adjusted geometric means comparing brain vs. plasma concentrations of voriconazole N-oxide. Natural-log transformed concentrations of voriconazole were analyzed using a mixed-effects model to obtain the adjusted mean difference (Test-Reference) and 90% confidence interval for the difference which were exponentiated to provide estimates of the ratio of the adjusted geometric means and 90% CI for the ratio; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; predose: ratio adjusted geometric means = 12.39, 90% CI [7.09 to 21.65] — Estimated value = ratio (%) of adjusted geometric means comparing brain (test) vs. plasma (reference) concentrations of voriconazole N-oxide
Statistical Analysis 2: Comparison: Voriconazole; Other estimated parameter represents the Day 3 post-dose ratio of the adjusted geometric means comparing brain vs. plasma concentrations of voriconazole N-oxide. Natural-log transformed concentrations of voriconazole were analyzed using a mixed-effects model to obtain the adjusted mean difference (Test-Reference) and 90% confidence interval for the difference which were exponentiated to provide estimates of the ratio of the adjusted geometric means and 90% CI for the ratio; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; postdose: ratio adjusted geometric means = 31.57, 90% CI [18.06 to 55.18] — [estimate comment as in outcome 3, analysis 1]

4. Primary Outcome: Brain Concentrations of N-oxide Metabolite
Description: Mean brain concentrations (ng/mL) of voriconazole N-oxide metabolite pre-dose and 2 hours post-dose measured by Fluorine (F) Magnetic Resonance Spectroscopy (F-MRS).
Time Frame: Day 3: pre-dose, 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Voriconazole
Number analyzed (Participants) | 12
ng/mL
  predose (Cmin) | 663.97 (677.55)
  2 hours postdose (C2h) | 1535.40 (1280.09)
Statistical Analysis 1: Comparison: Voriconazole; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; predose: ratio adjusted mean = 12.39, 90% CI [7.09 to 21.65] — Estimated value = ratio (%) of adjusted geometric means comparing brain (test) vs. plama (reference) concentrations of voriconazole N-oxide
Statistical Analysis 2: Comparison: Voriconazole; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; postdose: ratio adjusted mean = 31.57, 90% CI [18.06 to 55.18] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Arm/Group | Voriconazole
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=12)
Ear discomfort (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 1
Photophobia (Eye disorders) | 5
Vision blurred (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Head discomfort (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.